CLINICAL TRIAL: NCT05096416
Title: Three-dimensional (3D) Printed Hemodialysis Vascular Model for Increased Precision of Cannulation
Brief Title: Three-dimensional (3D) Printed Hemodialysis Vascular Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Michael Siedlecki, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022P000658
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Hemodialysis Access Failure
Keywords: hemodialysis; Magnetic resonance angiography; three-dimensional (3D) printed hemodialysis vascular model; Vascular access complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Control arm (No Intervention): Patients in this arm will have standard of care where they will be annulated by the palpation method by the dialysis technician and nurse.
- Intervention arm (Experimental): Patients in this arm will have a three-dimensional (3D) printed vascular access model to assist the dialysis technician and nurse in cannulation.
  Interventions: Device: The three-dimensional (3D) printed hemodialysis vascular model

INTERVENTIONS:
Device: The three-dimensional (3D) printed hemodialysis vascular model — The three-dimensional (3D) printed hemodialysis vascular model will be used as a guide map to cannulate the patients for hemodialysis and to minimize the risk of vascular access complications
  Arms: Intervention arm

SUMMARY:
Infiltration of a surgically-placed hemodialysis vascular access (HVA) is recognized as a major contributor to the high hospital re-admission rate in dialysis-dependent patients. Three dimensional modeling has been demonstrated as a critical tool for procedurists in preparation for surgical interventions but no such modeling is yet available for dialysis specialists to avoid the common complication of HVA infiltration. Contrast enhanced magnetic resonance angiography (MRA) can be used to generate a three dimensional image data that could render a three dimensional resin-based model of a vascular access.

DETAILED DESCRIPTION:
Hemodialysis is the most common treatment for End Stage Renal Disease (ESRD). For an optimal renal replacement therapy, a patent vascular access (VA) is essential. The importance of good vascular access maintenance has been strongly supported by the guidelines (1). Various hinderances render this goal unachievable. A well-known cause of VA failure is access infiltration, which is usually overlooked in clinical practices (2). The calculated economic burden attributable to VA complication is between $16,864 -US$20,961 and more than 50% is due to access infiltration alone (3). Imaging has a pivotal pre- and post-operative role in evaluating vascular access complications. Imaging modalities such as ultrasound (US), Digital Subtraction Angiography (DSA) and Magnetic Resonance Angiography (MRA) are available but their use is limited due to the limited view of plane available for visualization of vessel anatomy(4) and because of the deleterious side effects of the contrast agents used (5,6). Contrast enhanced Magnetic Resonance Angiography (MRA) provides an excellent means of imaging the vasculature (7) which can be reconstructed in a three- dimensional(3D) print. The skill set of dialysis technician nurses play a considerable role in achieving successful cannulation of the fistula. Due oftentimes to complicated vascular anatomy, cannulation based on cutaneous anatomic landmarks and physical examination can be deceiving. Even a minor error in cannulation can impair access longevity(3). The 3D image reconstruction provides a practical solution to generate a 3D VA model which can be used by the procedurists to cannulate the patients, reducing the complications and rate of re admissions. Overall, a significant reduction in the health care cost can be achieved

ELIGIBILITY:
Inclusion Criteria:

* Patients with a surgically placed hemodialysis access which has been used in the last 90 days or is being prepared for use in the next 90 days

Exclusion Criteria:

* Patients with only failed hemodialysis surgical access(es) that has/have not been used for >90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Quantify the number of dialysis treatments completed | 12 month

SECONDARY OUTCOMES:
Quantify the number of vascular access interventions over a 12-month period compared to controls | 12 month
Quantify annual hospitalization rate compared to controls | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Siedlecki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No